CLINICAL TRIAL: NCT02799914
Title: Evaluation of the Sinus-Venous Stent for the Treatment of Iliofemoral Venous Occlusive Disease: A Monocenter Post Market Clinical Follow-up Study
Brief Title: Evaluation of the Sinus-Venous Stent for the Treatment of Iliofemoral Venous Occlusive Disease
Status: Withdrawn | Type: Observational
Why Stopped: Difficult patient recruitment. No patients enrolled.
Sponsor: be Medical (Industry)
Collaborators: Archer Research (Industry)
Responsible Party: Sponsor
Other Study IDs: VS-01
Record Dates: First submitted 2015-12-07; First posted 2016-06-15 (Estimated); Last update posted 2019-02-08 (Actual); Status verified 2017-11

CONDITIONS: Venous Vascular Diseases and Syndromes
MeSH Terms: conditions — Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

INTERVENTIONS:
Device: Sinus-Venous stent (Optimed GmbH) — Stent implantation

SUMMARY:
Post market clinical follow-up study about the Sinus-venous stent. Patients with venous iliofemoral occlusive disease are treated with the Sinus-venous stent. This observational study will provide 1 year data about safety and efficacy.

ELIGIBILITY:
Inclusion Criteria:

1. Age at study entry is at least 18 years.
2. Patient must sign the informed consent form prior to the index-procedure.
3. Patient suffers from acute or chronic venous occlusive disease indicated to be treated with a venous stent.
4. Target lesion is located in the femoral vein, common femoral vein, external iliac vein, or common iliac vein.

Exclusion Criteria:

1. Intolerance to anticoagulant medication.
2. Contra-indication for prolonged anticoagulant treatment.
3. Life expectancy less than 1 year.
4. Target vessel has been stented before.
5. Coagulopathy or known uncorrectable bleeding diathesis.
6. Recent (<1 year) pulmonary embolism.
7. Pregnancy.
8. Known hypersensitivity to nitinol and/or nickel.
9. Known to be, or suspected of being unable to comply with the study protocol (e.g. no permanent address, known to be non-compliant or presenting an unstable psychiatric history).
10. Legal incapacity and/or other circumstances rendering the patient unable to understand the nature, scope and possible impact of the study.
11. Patients in custody by juridical order.
12. Patients who do not agree to the transmission of their coded data within the liability of documentation and notification.
13. Close affiliation with the investigational site: e.g. a close relative of the investigator or a possibly dependent person (e.g. employee or student of the investigational site).

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with venous iliofemoral occlusive disease.
Sampling Method: Non-Probability Sample
Enrollment: 0 (Actual)
Dates: Start 2016-04 (Actual); Primary Completion 2018-06 (Actual); Study Completion 2018-06 (Actual)

PRIMARY OUTCOMES:
Stent patency | 12 months
  Patency broken down in primary patency, assisted primary patency and secondary patency

SECONDARY OUTCOMES:
Technical success | Index-procedure (intraoperative)
  The index-procedure is the endovascular procedure in which the patient receives the device.
Revised venous clinical severity score | 12 months
Mortality | 12 months
Procedural complications | Index-procedure
Reintervention | 12 months
  Any peripheral venous intervention after the index-procedure to restore patency in the treated segment or outside the treated segment

CONTACTS AND LOCATIONS:
Overall Officials: Geert Lauwers, MD, Principal Investigator — Ziekenhuis Oost-Limburg
Locations (1):
- Ziekenhuis Oost-Limburg, Genk, Belgium

IPD SHARING:
Plan to Share IPD: No